CLINICAL TRIAL: NCT01304550
Title: Evaluation of the Accuracy of the Masimo Pulse-Hemoglobin-Meter Monitor in Surgical Patients
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200917394; 200917394-1
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Accuracy of Non-invasive Hemoglobin Monitor
Keywords: non-invasive; hemoglobin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective comparison of hemoglobin measurements obtained by arterial blood gas analysis and the Masimo Continuous Hemoglobin Monitor

DETAILED DESCRIPTION:
The chief objective of this study is to internally validate the accuracy of the Masimo SpHb (TM) technology as compared to our laboratory measurement of Hb. We have been using the Masimo SpHb monitor on patients who underwent open heart surgery, hepatic resection, kidney transplant and aortic aneurysm repair since January 2009. These patients also had hemoglobin concentration measurements as part of the arterial blood gas analysis performed by our laboratory to evaluate intraoperative ventilation and electrolyte changes. We will collate the laboratory measurements with the Masimo SpHb values documented in the anesthetic records.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had indwelling arterial catheters placed for surgeries that involved major blood loss and who had serial hemoglobin concentration measurements for their surgeries, since January 2009. This will represent approximately 50 patients.

Exclusion Criteria:

* Inclusion criteria are patients undergoing major surgery from January 2009 - April 2009, who had continuous hemoglobin pulse oximetry readings form the Masimo SpHb monitor and serial hemoglobin concentration measurement from the lab. Patient who did not have these studies will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patience undergoing elect cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of Masimo Monitor | 1 Year
  365 Days

CONTACTS AND LOCATIONS:
Overall Officials: Neal W. Fleming, M.D., Ph.D., Study Director — Director, Cardiovascular and Thoracic Anesthesiology, UC Davis, Department of Anesthesiology and Pain Medicine; Aubrey Yao, M.D., Principal Investigator — Faculty, Cardiovascular and Thoracic Anesthesiology, UC Davis, Department of Anesthesiology and Pain Medicine; Gudrun Kungys, M.D., Principal Investigator — Faculty, Cardiovascular and Thoracic Anesthesiology, UC Davis, Department of Anesthesiology and Pain Medicine